CLINICAL TRIAL: NCT05900453
Title: Novel Strategies for Personalized Clinical Decisions in Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: ATI Physical Therapy (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-1246
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Total Knee Replacement
Keywords: precision medicine; prognosis; patient-centered care; Decision Support Systems, Clinical
MeSH Terms: interventions — Compact Disks; Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care TKA rehabilitation: This cohort of patients received Usual Care TKA rehabilitation at two outpatient physical therapy clinics in the Greenville, South Carolina, USA area. These patients received treatment guided by their clinician's professional judgment and the clinic's best practice guidelines for TKA.
- CDS tool TKA rehabilitation: This cohort of patients received TKA rehabilitation at the same two outpatient physical therapy clinics in the Greenville, South Carolina, USA area. These patients also received treatment guided by their clinician's professional judgement and the clinic's best practice guidelines. Additionally, this cohort of patients was exposed to the CDS tool (i.e., clinicians used the tool to view personalized information about the patient at least once during the patient's episode of care).
  Interventions: Other: Clinical decision support (CDS) tool

INTERVENTIONS:
Other: Clinical decision support (CDS) tool — The web-based clinical decision support (CDS) tool uses patient information (e.g., age, sex, BMI, perioperative status) to create personalized predictions of recovery following knee replacement. The CDS tool predicts range of motion, physical function, and pain recovery. Clinicians can use these predictions to (1) inform patients of their expected prognosis, (2) monitor patients' recovery against their predicted recovery, and (3) tailor treatments according to individual patients' needs.
  Clinicians were provided with basic training for how to use the CDS tool, and were given examples of how to integrate it into clinical care. However, the CDS tool did not dictate any treatment decisions; clinicians were free to use the CDS tool at their discretion to inform decision making.
  Groups: CDS tool TKA rehabilitation

SUMMARY:
This study will compare the postoperative recovery of two patient cohorts who attended outpatient physical therapy at two clinics in the Greenville, South Carolina area. The Usual Care cohort received care according to each clinic's pre-existing care guidelines. The CDS Cohort received care informed by a new clinical decision support (CDS) tool.

DETAILED DESCRIPTION:
In this cohort study, the investigators will use regression to examine whether CDS tool exposure was associated with patient outcomes after total knee replacement. Linear mixed effect models will be used for continuous outcomes that have multiple assessment points per patient. For count outcomes (e.g., visit utilization), the investigators will use Poisson/negative binomial regression or linear regression with appropriate outcome transformations.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent TKA for primary knee osteoarthritis
* Patient underwent postoperative TKA rehabilitation at one of the two participating physical therapy clinics in the Greenville, SC area

Exclusion Criteria:

* Patients < 40 years old
* Patients whose total episode of care length in outpatient physical therapy was < 21 days
* Patients who attended < 3 outpatient physical therapy visits throughout their episode of care
* Outcomes collected > 6 months after surgery (except for visit utilization, which can include data up to 1 year after surgery)
* Patients who were not exposed to the CDS tool, but were treated by a clinician who was trained to use the CDS tool

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend post-TKA rehabilitation at the participating outpatient physical therapy clinics in the Greenville, SC area.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS-JR) | KOOS-JR was assessed postoperatively up to 6 months after surgery
  The KOOS-JR is a patient-reported measure of physical function developed specifically for patients with total knee arthroplasty (TKA). The KOOS-JR is scored on a 100-point scale with 0 representing complete knee disability and 100 representing perfect knee health. It can be completed quickly (only 7 items) and has established validity, reliability, and responsiveness in the TKA population.

SECONDARY OUTCOMES:
Outpatient Physical Therapy Visit Utilization | All visits from initial evaluation to discharge up to 1 year after surgery
  The total number of outpatient physical therapy visits attended by each patient during the year immediately following their TKA will be extracted from the electronic medical record. Only visits associated with the patient's episode of care for TKA will be included.
Time Up and Go (TUG) | TUG was assessed postoperatively up to 6 months after surgery
  The TUG is a basic measure of mobility and balance that consists of rising from a seated position, walking three meters, and pivoting and returning to the original seated position. The TUG is responsive to change with adequate reliability in the acute recovery period after TKA.
Surveys of patients' perceived knowledge of their recovery and engagement in their rehabilitation. | Surveys were assessed postoperatively up to 6 months after surgery
  Patients completed surveys regarding their perceived knowledge of their postoperative recovery and their engagement in rehabilitation decision making. The surveys were scored on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).
Knee range of motion (ROM) | ROM was assessed postoperatively up to 6 months after surgery
  Knee flexion and extension ROM was measured manually by goniometry, which is a valid and reliable technique for measuring knee mobility. Recovery of ROM after TKA is necessary for many functional activities and is emphasized in rehabilitation after TKA.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Stevens-Lapsley, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- ATI Physical Therapy, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No